CLINICAL TRIAL: NCT02669784
Title: Does Reduction in Contrast Administration Dose in Computed Tomography Arteriograms Degrade Image Quality? A Single Institutional Review of an Ultra-low Contrast Dose Protocol
Brief Title: Computed Tomography Arteriograms (CTA) Volume Dose Reduction Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Rekha Cherian, Physician, Milton S. Hershey Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 3932
Record Dates: First submitted 2016-01-21; First posted 2016-02-01 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Aortic Aneurysm; Contrast Induced Nephropathy; Aortic and Arterial Anomalies
MeSH Terms: conditions — Aortic Aneurysm | interventions — Contrast Media; Iohexol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Dose Contrast (40mL) (Active Comparator): CTA of the chest: 40 mL of intravenous contrast at a rate of 5mL/sec. A region of interest (ROI) to trigger the scan will be placed in the aortic arch. If scan is performed using high pitch helical mode, the scan delay will be increased by 2 seconds. The Low Dose scan will then be compared to the standard of care high dose scan of the same area taken at a previous date.
  Interventions: Drug: Low Dose Contrast (Omnipaque) 40mL
- Low Dose Contrast (50mL) (Active Comparator): CTA of the abdomen OR or CTA of the chest and abdomen or CTA of the abdomen and pelvis or CTA of the chest, abdomen and pelvis: 50 mL of intravenous contrast at a rate 5mL/sec. A region of interest (ROI) to trigger the scan will be placed in the aortic arch. If scan is performed using high pitch helical mode, the scan delay will be increased by 2 seconds. The Low Dose scan will then be compared to the standard of care high dose scan of the same area taken at a previous date.
  Interventions: Drug: Low Dose Contrast (Omnipaque) 50 mL

INTERVENTIONS:
Drug: Low Dose Contrast (Omnipaque) 40mL — The patient will be administered a low dose, 40mL of intravenous contrast (Omnipaque) at a rate of 5mL/sec based on the area of the body being scanned (chest versus chest and abdomen versus chest, abdomen and pelvis). This will be compared to the patient's prior examination performed with 100mL of intravenous contrast at a rate of 4mL/sec.
  Arms: Low Dose Contrast (40mL)
Drug: Low Dose Contrast (Omnipaque) 50 mL — The patient will be administered a low dose, 50mL of intravenous contrast (Omnipaque) at a rate of 5mL/sec based on the area of the body being scanned (chest versus chest and abdomen versus chest, abdomen and pelvis). This will be compared to the patient's prior examination performed with 100mL of intravenous contrast at a rate of 4mL/sec.
  Arms: Low Dose Contrast (50mL)

SUMMARY:
The purpose of the study is to determine if the dose of contrast (Omnipaque) administered for Computed Tomography Arteriograms (CTA) can be reduced without degradation of image quality. The hypothesis is that there is no difference in image quality using ultra-low dose contrast in CTA exams compared to routine, standard of care dose exams.

DETAILED DESCRIPTION:
Any adult patient age 18 and above, scheduled for routine CTA (Computed Tomography Arteriograms) of the chest or chest, abdomen and pelvis meeting inclusion criteria and not meeting any exclusion criteria will be included in the study. The patient will be administered a low dose of intravenous contrast based on the study examination as described below.

CTA of the chest: 40 mL of intravenous contrast (Omnipaque) at a rate of 5mL/sec. A region of interest (ROI) to trigger the scan will be placed in the aortic arch. If scan is performed using high pitch helical mode, the scan delay will be increased by 2 seconds.

CTA of the chest and abdomen or CTA of the chest, abdomen and pelvis: 50 mL of intravenous contrast (Omnipaque) at a rate 5mL/sec. A region of interest (ROI) to trigger the scan will be placed in the aortic arch. If scan is performed using high pitch helical mode, the scan delay will be increased by 2 seconds.

Following the examination, the primary investigator (PI) or team members will evaluate the images obtained with low contrast dose and each patient's prior CTA examination performed with routine contrast dose, 100mL at a rate of 4mL/sec. This will be done by quantitative and qualitative measures. For the quantitative portion, the PI or team members will place regions of interest on predetermined arterial locations to obtain measure the degree of opacification. For qualitative measurement, the images will be presented in a blind fashion to two thoracic trained board certified radiologists and a board certified interventional radiologist to determine the quality of the images based on a Likert numerical scale. Qualitative and quantitative data for the images obtained with low contrast dose and those for the prior CTA examinations performed with routine contrast dose will be compared. This data along with details of the scan protocol (dose, dose rate, scanning parameters etc.) and demographic data (such as sex, age and BMI at the time of examination) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient scheduled for a computed tomographic arteriogram (CTA) of the chest or chest, abdomen and pelvis who had undergone a prior CTA performed with the standard contrast dose (100 mL) at this institution will be included in the study
* The follow-up scan will be routine standard of care, no emergency imaging patient will be approached for this research

Exclusion Criteria:

* Patients with no prior CTA imaging for comparison
* Any pediatric patient (age <18)
* BMI >40
* Inability to follow instructions
* Allergy to intravenous contrast
* GFR less than 30 mL/min/1.73 m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Seehofnerova A, Kok M, Mihl C, Douwes D, Sailer A, Nijssen E, de Haan MJ, Wildberger JE, Das M. Feasibility of low contrast media volume in CT angiography of the aorta. Eur J Radiol Open. 2015 Apr 28;2:58-65. doi: 10.1016/j.ejro.2015.03.001. eCollection 2015. PMID 26937437
- [Background] Rubin GD. MDCT imaging of the aorta and peripheral vessels. Eur J Radiol. 2003 Mar;45 Suppl 1:S42-9. doi: 10.1016/s0720-048x(03)00036-6. PMID 12598026
- [Background] Gleeson TG, Bulugahapitiya S. Contrast-induced nephropathy. AJR Am J Roentgenol. 2004 Dec;183(6):1673-89. doi: 10.2214/ajr.183.6.01831673. No abstract available. PMID 15547209
- [Background] Vanommeslaeghe F, De Mulder E, Van de Bruaene C, Van de Bruaene L, Lameire N, Van Biesen W. Selecting a strategy for prevention of contrast-induced nephropathy in clinical practice: an evaluation of different clinical practice guidelines using the AGREE tool. Nephrol Dial Transplant. 2015 Aug;30(8):1300-6. doi: 10.1093/ndt/gfv220. Epub 2015 Jun 4. PMID 26047631
- [Background] Meschi M, Detrenis S, Musini S, Strada E, Savazzi G. Facts and fallacies concerning the prevention of contrast medium-induced nephropathy. Crit Care Med. 2006 Aug;34(8):2060-8. doi: 10.1097/01.CCM.0000227651.73500.BA. PMID 16763513
- [Background] Walsh SR, Tang T, Gaunt ME, Boyle JR. Contrast-induced nephropathy. J Endovasc Ther. 2007 Feb;14(1):92-100. doi: 10.1583/06-2035.1. PMID 17291156
- [Background] Gussenhoven MJ, Ravensbergen J, van Bockel JH, Feuth JD, Aarts JC. Renal dysfunction after angiography; a risk factor analysis in patients with peripheral vascular disease. J Cardiovasc Surg (Torino). 1991 Jan-Feb;32(1):81-6. PMID 2010458
- [Background] Diehm N, Pena C, Benenati JF, Tsoukas AI, Katzen BT. Adequacy of an early arterial phase low-volume contrast protocol in 64-detector computed tomography angiography for aortoiliac aneurysms. J Vasc Surg. 2008 Mar;47(3):492-8. doi: 10.1016/j.jvs.2007.11.004. PMID 18295101
- [Background] Viteri-Ramirez G, Garcia-Lallana A, Simon-Yarza I, Broncano J, Ferreira M, Pueyo JC, Villanueva A, Bastarrika G. Low radiation and low-contrast dose pulmonary CT angiography: Comparison of 80 kVp/60 ml and 100 kVp/80 ml protocols. Clin Radiol. 2012 Sep;67(9):833-9. doi: 10.1016/j.crad.2011.11.016. Epub 2012 Jun 8. PMID 22683247
- [Background] Wu CC, Lee EW, Suh RD, Levine BS, Barack BM. Pulmonary 64-MDCT angiography with 30 mL of IV contrast material: vascular enhancement and image quality. AJR Am J Roentgenol. 2012 Dec;199(6):1247-51. doi: 10.2214/AJR.12.8739. PMID 23169715

RESULTS

PARTICIPANT FLOW:
Groups:
- Contrast (Omnipaque) Low Dose (40mL): CTA of the chest: 40 mL of intravenous contrast (omnipaque) at a rate of 5mL/sec. A region of interest (ROI) to trigger the scan will be placed in the aortic arch. If scan is performed using high pitch helical mode, the scan delay will be increased by 2 seconds.
  This will be compared to the patient's prior examination performed with 100 mL of intravenous contrast.
- Contrast (Omnipaque) Low Dose (50mL): CTA of the chest and abdomen or CTA of the chest, abdomen and pelvis: 50 mL of intravenous contrast at a rate 5mL/sec. A region of interest (ROI) to trigger the scan will be placed in the aortic arch. If scan is performed using high pitch helical mode, the scan delay will be increased by 2 seconds.
  This will be compared to the patient's prior examination performed with 100 mL of intravenous contrast.
Period: Overall Study
Arm/Group | Contrast (Omnipaque) Low Dose (40mL) | Contrast (Omnipaque) Low Dose (50mL)
Started | 18 | 16
Completed | 18 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Contrast (40mL) | Low Dose Contrast (50mL) | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 11 | 10 | 21
Age, Continuous [Mean (Full Range); unit: years] | 66 [55 to 85] | 62 [20 to 86] | 66 [20 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 12 | 11 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 18 | 16 | 34
Type of Scan [Count of Participants; unit: Participants]
  Chest Scan | 17 | 0 | 17
  Abdomen Scan | 1 | 0 | 1
  Abdomen and Pelvis Scan | 0 | 4 | 4
  Chest, Abdomen, and Pelvis Scan | 0 | 11 | 11
  Chest and Abdomen Scan | 0 | 1 | 1
Contrast, 100mL: Scan Dose [Count of Participants; unit: Participants] | 18 | 16 | 34
Contrast, 100mL: Ascending: Sinotubular Junction Measurement [Mean (Full Range); unit: hounsfield units] | 317.5 [240.5 to 434.4] | 397.6 [269.5 to 690.3] | 352.6 [240.5 to 690.3]
Contrast, 100mL: Descending: Pulmonary Artery Measurement [Mean (Full Range); unit: hounsfield units] | 283.9 [215.8 to 427.8] | 338.1 [244.3 to 560.5] | 329 [215.8 to 560.5]
Contrast, 100mL: Celiac Measurement [Mean (Full Range); unit: hounsfield units] | 309.1 [214.7 to 444.7] | 363.8 [212.8 to 696.6] | 334.2 [212.8 to 696.6]
Contrast, 100mL: Bifurcation Measurement [Mean (Full Range); unit: hounsfield units] | 322.4 [256.2 to 395.9] | 361.4 [226.3 to 566.3] | 354.9 [226.3 to 566.3]
Contrast, 100mL: Right Common Femoral Measurement [Mean (Full Range); unit: hounsfield units] | 331.3 [301.8 to 360.8] | 331 [147.9 to 615.3] | 331 [147.9 to 615.3]
Contrast, 100mL: Left Common Femoral Measurement [Mean (Full Range); unit: hounsfield units] | 332 [289.4 to 374.7] | 350.9 [206 to 490] | 348.5 [206 to 490]
Contrast, 100mL: CTA Vessel Opacification Grading 1 [Mean (Full Range); unit: score on a scale] — 5 Point Grading Scale was used to determine CTA Vessel Opacification by a Board Certified Radiologist.
  1. Poor opacification with no difference in attenuation of the lumen compared to the wall of the vessel. Non diagnostic.
  2. Decreased opacification. Little to no difference in attenuation between the lumen and the wall. Non diagnostic.
  3. Moderate opacification of the lumen of the vessel. Diagnostic study.
  4. Good opacification of the lumen of the vessel.
  5. Excellent opacification of the lumen of the vessel with distinct difference in attenuation of the wall and lumen of the vessel.
  score on a scale | 4.9 [4 to 5] | 4.7 [4 to 5] | 4.79 [4 to 5]
Contrast, 100mL: CTA Vessel Opacification Grading 2 [Mean (Full Range); unit: score on a scale] — 5 Point Grading Scale was used to determine CTA Vessel Opacification by a second Board Certified Radiologist.
  1. Poor opacification with no difference in attenuation of the lumen compared to the wall of the vessel. Non diagnostic.
  2. Decreased opacification. Little to no difference in attenuation between the lumen and the wall. Non diagnostic.
  3. Moderate opacification of the lumen of the vessel. Diagnostic
  4. Good opacification of the lumen of the vessel.
  5. Excellent opacification of the lumen of the vessel with distinct difference in attenuation of the wall and lumen of the vessel.
  score on a scale | 4.8 [4 to 5] | 4.8 [4 to 5] | 4.8 [4 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Ascending Sinotubular Junction Measurement
Description: Following image acquisition, quantitative analysis was performed by measurement of the attenuation of the contrast bolus by use of Hounsfield Units. Measurement was taken at the ascending aorta near the sinotubular junction.
Time Frame: At 30 days
Population: Ascending Sinotubular Junction Measurement was assessed for the following scans: Chest, Abdomen & Pelvis, and Chest, Abdomen, & Pelvis
Measure: Mean (Full Range); unit: Hounsfield units
Arm/Group | Contrast (Omnipaque) Low Dose (40mL) | Contrast (Omnipaque) Low Dose (50mL)
Number analyzed (Participants) | 17 | 10
Hounsfield units | 246.4 [135 to 460.3] | 287.5 [125 to 443.13]

2. Primary Outcome: Descending Thoracic Aorta Measurement
Description: Following image acquisition, quantitative analysis was performed by measurement of the attenuation of the contrast bolus by use of Hounsfield Units. A measurement was taken from the distal abdominal aorta prior to the bifurcation.
Time Frame: 30 days
Population: Descending Thoracic Aorta Measurement was assessed for the following scans: Chest, and Chest, Abdomen, & Pelvis
Measure: Mean (Full Range); unit: Hounsfield units
Arm/Group | Contrast (Omnipaque) Low Dose (40mL) | Contrast (Omnipaque) Low Dose (50mL)
Number analyzed (Participants) | 17 | 10
Hounsfield units | 261.9 [119.4 to 452.8] | 312.8 [185.3 to 494.3]

3. Primary Outcome: Celiac Measurement
Description: Following image acquisition, quantitative analysis was performed by measurement of the attenuation of the contrast bolus by use of Hounsfield Units. A measurement was taken from the proximal abdominal aorta at the level of the celiac axis.
Time Frame: 30 days
Population: Celiac Measurement was assessed for all scans: Chest, Abdomen, Abdomen & Pelvis, and Chest, Abdomen, & Pelvis.
Measure: Mean (Full Range); unit: Hounsfield units
Arm/Group | Contrast (Omnipaque) Low Dose (40mL) | Contrast (Omnipaque) Low Dose (50mL)
Number analyzed (Participants) | 18 | 16
Hounsfield units | 243.8 [115.9 to 453.3] | 329.5 [146.2 to 813.0]

4. Primary Outcome: Burfication Measurement
Description: as for outcome 2
Time Frame: 30 days
Population: Burfication measurements were taken from the following scans: Abdomen, Abdomen & Pelvis, and Chest, Abdomen, & Pelvis.
Measure: Mean (Full Range); unit: Hounsfield units
Arm/Group | Contrast (Omnipaque) Low Dose (40mL) | Contrast (Omnipaque) Low Dose (50mL)
Number analyzed (Participants) | 1 | 16
Hounsfield units | 336.2 [NA to NA] — Only 1 participant was analyzed therefore a full range cannot be calculated. | 321.2 [126.4 to 581.0]

5. Primary Outcome: Right Common Femoral Artery Measurement
Description: Following image acquisition, quantitative analysis was performed by measurement of the attenuation of the contrast bolus by use of Hounsfield Units. A measurement was taken from the right common femoral artery.
Time Frame: 30 days
Population: All participants in the Contrast (Omnipaque) Low dose (40mL) underwent only a CTA of the chest or abdomen which is incapable of measuring the right common femoral artery.
Measure: Mean (Full Range); unit: Hounsfield units
Arm/Group | Contrast (Omnipaque) Low Dose (40mL) | Contrast (Omnipaque) Low Dose (50mL)
Number analyzed (Participants) | 0 | 14
Hounsfield units |  | 314.5 [168.9 to 588.5]

6. Primary Outcome: Left Common Femoral Artery Measurement
Description: as for outcome 5
Time Frame: 30 days
Population: All participants in the Contrast (Omnipaque) Low dose (40mL) underwent only a CTA of the chest or abdomen which is incapable of measuring the Left common femoral artery
Measure: Mean (Full Range); unit: Hounsfield units
Arm/Group | Contrast (Omnipaque) Low Dose (40mL) | Contrast (Omnipaque) Low Dose (50mL)
Number analyzed (Participants) | 0 | 14
Hounsfield units |  | 309.5 [143.8 to 561.0]

7. Primary Outcome: CTA Vessel Opacification Grading 1
Description: 5 Point Grading Scale was used to determine CTA Vessel Opacification by a Board Certified Radiologist.
  1. Poor opacification with no difference in attenuation of the lumen compared to the wall of the vessel. Non diagnostic.
  2. Decreased opacification. Little to no difference in attenuation between the lumen and the wall. Non diagnostic.
  3. Moderate opacification of the lumen of the vessel. Diagnostic study.
  4. Good opacification of the lumen of the vessel.
  5. Excellent opacification of the lumen of the vessel with distinct difference in attenuation of the wall and lumen of the vessel.
Time Frame: 30 days
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Contrast (Omnipaque) Low Dose (40mL) | Contrast (Omnipaque) Low Dose (50mL)
Number analyzed (Participants) | 18 | 16
score on a scale | 4 [2 to 5] | 4.3 [3 to 5]

8. Primary Outcome: CTA Vessel Opacification Grading 2
Description: 5 Point Grading Scale was used to determine CTA Vessel Opacification by a second Board Certified Radiologist.
  1. Poor opacification with no difference in attenuation of the lumen compared to the wall of the vessel. Non diagnostic.
  2. Decreased opacification. Little to no difference in attenuation between the lumen and the wall. Non diagnostic.
  3. Moderate opacification of the lumen of the vessel. Diagnostic
  4. Good opacification of the lumen of the vessel.
  5. Excellent opacification of the lumen of the vessel with distinct difference in attenuation of the wall and lumen of the vessel.
Time Frame: 30 days
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Contrast (Omnipaque) Low Dose (40mL) | Contrast (Omnipaque) Low Dose (50mL)
Number analyzed (Participants) | 18 | 16
score on a scale | 4.2 [3 to 5] | 4.4 [3 to 5]

ADVERSE EVENTS:
Time Frame: 30 days
Groups:
- Low Dose Contrast (40mL): CTA of the chest: 40 mL of intravenous contrast (omnipaque) at a rate of 5mL/sec. A region of interest (ROI) to trigger the scan will be placed in the aortic arch. If scan is performed using high pitch helical mode, the scan delay will be increased by 2 seconds. . The Low Dose scan will then be compared to the standard of care high dose scan of the same area taken at a previous date.
- Low Dose Contrast (50mL): CTA of the chest and abdomen or CTA of the chest, abdomen and pelvis: 50 mL of intravenous contrast at a rate 5mL/sec. A region of interest (ROI) to trigger the scan will be placed in the aortic arch. If scan is performed using high pitch helical mode, the scan delay will be increased by 2 seconds. The Low Dose scan will then be compared to the standard of care high dose scan of the same area taken at a previous date.
Arm/Group | Low Dose Contrast (40mL) | Low Dose Contrast (50mL)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 0/18 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-16): https://cdn.clinicaltrials.gov/large-docs/84/NCT02669784/Prot_SAP_000.pdf